CLINICAL TRIAL: NCT04315532
Title: Relationship of Sex Steroid and Stress Markers in Saliva and Gingival Crevicular Fluid With Pregnancy
Brief Title: The Effect of Periodontal Treatment on Stress and Pregnancy Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ozge Gokturk, Principal Investigator, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018.06.05.1298
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy Gingivitis
Keywords: Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnancy Group (Active Comparator): GCF and saliva samples were taken from pregnant gingivitis patients before treatment and after 8 weeks. GCF and saliva samples were taken from pregnant periodontal healty individuals baseline and after 8 weeks.
  Intervention: Non-surgical periodontal treatment was performed for pregnant gingivitis patients. Gingival crevicular fluid (GCF) and saliva samples were taken.
  Interventions: Other: Non-surgical periodontal treatment; Other: Saliva samples; Other: GCF samples
- Non-Pregnancy Group (Active Comparator): GCF and saliva samples were taken from non-pregnant gingivitis patients before treatment and after 8 weeks. GCF and saliva samples were taken from periodontal healty individuals baseline and after 8 weeks.
  Intervention: Non-surgical periodontal treatment was performed for non-pregnant gingivitis patients. Gingival crevicular fluid (GCF) and saliva samples were taken.
  Interventions: Other: Non-surgical periodontal treatment; Other: Saliva samples; Other: GCF samples

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Non-surgical periodontal treatment was performed for pregnant and non-pregnant gingivitis patients. Gingival crevicular fluid (GCF) and saliva samples were taken from all patients baseline and after 8 weeks.
Other: Saliva samples — Saliva samples were taken from patients for the evaluation of sex steroid and stress markers baseline and after 8 weeks.
Other: GCF samples — GCF samples were taken from patients for the evaluation of stress markers baseline and after 8 weeks.

SUMMARY:
There is a relationship between stress and pregnancy gingivitis. This relationship may be double-sided.

DETAILED DESCRIPTION:
The aim of this clinical study was to determine the effect of non-surgical mechanical periodontal treatment on sex steroid and stress markers at pregnancy gingivitis. A total of 84 subjects; 22 pregnant women with gingivitis (group 1) and 25 pregnant women with periodontal healthy (pregnant group), group 2), 22 non-pregnant women with gingivitis (group 3) and 15 non-pregnant women with periodontal healthy (non-pregnant group), group 4) participated in this study. Clinically, plaque index, gingival index, and probing pocket depth were measured at baseline and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 24-50
* being pregnant for 23-30 weeks (for pregnant individuals)
* not smoking.

Exclusion Criteria:

* using antimicrobial or anti-inflammatory therapy within the previous 3 months,
* having systemic disease,
* having periodontitis,
* having deep caries lesions, and remnant roots and
* having lactation

Ages: 24 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Dehydroepiandrosterone (DHEA) | Baseline and after 8 weeks
  The changes in DHEA levels within 8 weeks. Higher values represent a worse outcome. The decrease in DHEA levels is expected after periodontal treatment.
estrogen | Baseline and after 8 weeks
  The changes in estrogen levels within 8 weeks. Higher values represent a worse outcome. The decrease in estrogen levels is expected after periodontal treatment.

SECONDARY OUTCOMES:
Gingival index | Baseline and after 8 weeks
  The changes in gingival index level after periodontal treatment. Gingival index was measured for determining the severity of disease and clinical outcome. Higher values represent a worse outcome. After periodontal treatment, a reduction in gingival index value is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Gokturk, Principal Investigator — Abant Izzet Baysal